CLINICAL TRIAL: NCT05142826
Title: Investigation of Strategies to Reduce the Impact of the Relative Age Effect in Kindergarten
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: University at Buffalo (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-20-0389; R34MH122212 (NIH)
Record Dates: First submitted 2021-11-08; First posted 2021-12-03 (Actual); Results first posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; kindergarten; relative age effect
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Schools

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Observers are masked to group assignment of the participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- School as Usual (Active Comparator): School procedures as typically used and implemented.
  Interventions: Other: School as Usual
- Immediate Relative Age Effect Intervention (Experimental): Relative age effect intervention administered in the Fall in school.
  Interventions: Behavioral: Relative Age Effect Intervention
- Delayed Relative Age Effect Intervention (Experimental): Relative age effect intervention administered after the Winter break in school.
  Interventions: Behavioral: Relative Age Effect Intervention

INTERVENTIONS:
Behavioral: Relative Age Effect Intervention — School-based consultation to establish a developmentally appropriate daily behavior report; teacher education regarding developmentally appropriate behaviors; teacher consultation to promote positive behavior supports.
  Arms: Delayed Relative Age Effect Intervention; Immediate Relative Age Effect Intervention
Other: School as Usual — Interventions and supports as provided through usual care
  Arms: School as Usual

SUMMARY:
There is now clear evidence that children entering kindergarten, that are relatively young for the grade (e.g., born in the months immediately preceding the school entry cut-off) are at significantly more risk for receiving an ADHD diagnosis and being prescribed stimulant medication. These risks appear to be related solely to age of entry when other explanatory variables are controlled. This situation, termed the "Relative Age Effect"has potentially serious consequences for kindergarten children (e.g., greater likelihood of being prescribed psychoactive medication to control behavior).

The present proposal aims to develop a teacher intervention to attenuate the impact of the relative age effect on young kindergarteners with elevated ADHD symptoms, and test the correspondence between the hypothesized mechanisms and treatment outcomes related to ADHD (e.g., symptoms, impairment). Following intervention development and refinement, 60 children entering kindergarten in the fall, and young for the grade, will be randomly assigned to (1) Kindergarten as Usual (KAU); (2) a Relative Age Effect prevention intervention administered immediately; or (3) a Relative Age Effect prevention intervention administered mid-year. In the intervention groups, teachers will be introduced to the relative age effect, receive information on how to anchor behavioral ratings in developmental norms, and implement a positive behavioral support to support growth in the child across the kindergarten school year.

Primary aims will be to demonstrate the feasibility and acceptability of the intervention approach as well as the ability of the team to retain young children in a longitudinal trial. Further, the hypothesized mechanisms (e.g., improved neurocognitive functioning; improved teacher use of positive behavioral supports) will be measured and correspondence to hypothesized outcomes (e.g., reduced ADHD symptoms and impairment) will be evaluated. Anticipated benefits include attenuation of any negative effects for children who receive intervention, and risks include breach of confidentiality and worsening of symptoms initially if an intervention is instituted. The knowledge to be gained is important as it could reduce untoward outcomes for the relatively youngest children in the grade.

DETAILED DESCRIPTION:
The entry to kindergarten is one of the most memorable and important milestones in a child's school career. Positive and quality kindergarten experiences have been associated with meaningful outcomes sustained into adulthood including greater rates of college attendance/higher earnings. Kindergarten entry is one of the first educational transitions made by a family, and it may cause stress and present new challenges for children and families. Given the increased demands that are associated with school entry and the concerns parents may have about this developmental milestone, there are numerous popular press and policy recommendations (e.g., National Association for the Education of Young Children), as well as empirical papers, that weigh in on the appropriate age to start kindergarten.

The transition to kindergarten is of particular concern for parents of children with ADHD, especially those relatively young for the grade. There is converging evidence suggesting that children who are young for their kindergarten class (e.g., they have a birthdate that falls within the months immediately preceding the cut-off date, typically August through November) are at increased risk for a range of negative educational outcomes including lower academic achievement, grade retention, social impairments, and ADHD diagnosis . These risks appear to be related to age of entry when other explanatory variables are controlled. Thus, these studies suggest that the robust evidence that children closest to an arbitrary cut-off date are disproportionally at-risk for negative social, behavioral, and educational outcomes is solely a consequence of educational policy - a phenomenon called the Relative Age Effect (RAE). Together, the consequence of these risks are 1.5x increased ADHD diagnostic rates and increased ADHD treatment with psychoactive medication for children relatively younger for their kindergarten grade .

There are prominent, candidate mechanisms that may explain the differential risk for children with ADHD who are also young for the grade. First, if a teacher is basing behavioral expectations for children in the classroom based on the relatively older children in the class, children who are relatively younger and have behaviors that are attributed to having considerable delays, even in situations where the child is acting in a manner consistent with their chronological age. Over time, if teachers are issuing frequent commands/reprimands, a coercive process may develop. Second, given expected variability in neurocognitive processing at this age level, inappropriate demands may fail to facilitate, and potentially even slow, the development of executive functions. The present proposal aims to reduce functional impairments and ADHD symptom levels by investigating whether evidence-based school treatment for ADHD (e.g., positive behavior supports) coupled with teacher training on the RAE results in improved school functioning for children with elevated ADHD symptoms prior to the kindergarten year. Further, the potential mechanism for the impairment experienced by children with ADHD will be explored, by investigating whether the impairments are due to characteristics of the child (e.g., deficits in neurocognitive development), the classroom (e.g., teacher classroom management strategies), or both.

ELIGIBILITY:
Inclusion Criteria:

* enrolling in Kindergarten
* has a date of birth 4 months prior to the respective state cut-off for school entry
* does not have an Individualized Education program for behavioral concerns
* has not been retained in school or "red-shirted" by parents.

Exclusion Criteria:

* outside of the targeted birthdate range
* diagnosed with autism, psychosis, or disruptive mood dysregulation disorder
* taking psychoactive medication for mood, behavior, or inattention,
* in a classroom with an already enrolled study participant.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Children and Families, Amherst, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified, anonymous data will be shared for the main outcome measures of the Disruptive Behavior Disorders Rating Scale and Impairment Rating Scale
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Six months after the completion of the project.
Access Criteria: Data will be shared through the NIMH data-sharing repository.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | School as Usual | Immediate Relative Age Effect Intervention | Delayed Relative Age Effect Intervention
Started | 20 | 21 | 21
Completed | 9 | 16 | 14
Not Completed | 11 | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | School as Usual | Immediate Relative Age Effect Intervention | Delayed Relative Age Effect Intervention | Total
Number analyzed (Participants) | 20 | 21 | 21 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 21 | 21 | 62
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 13 | 28
  Male | 13 | 13 | 8 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 6 | 11
  White | 9 | 15 | 10 | 34
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 8 | 2 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Disruptive Behavior Disorders Rating Scale
Description: Average score for ADHD symptom ratings on the Disruptive Behavior Disorders rating scale Average score ranges from 0.0 to 3.0 with higher scores indicating greater impairment.
Time Frame: Baseline (Fall), 3 Months (Winter), 6 Months (Spring) and 12 Months (First Grade Follow-up)
Measure: Mean (Standard Deviation); unit: score on the scale
Arm/Group | School as Usual | Immediate Relative Age Effect Intervention | Delayed Relative Age Effect Intervention
Number analyzed (Participants) | 20 | 21 | 21
score on the scale
  Baseline Fall Assessment | .8 (.51) | 1.12 (.8) | 1.03 (.72)
  Winter Assessment | 1.33 (.83) | 1.15 (.70) | 1.28 (.85)
  Spring Assessment | 1.34 (.91) | 1.13 (.80) | 1.00 (.65)
  First Grade Follow-up | 1.19 (.58) | 1.12 (.83) | 1.05 (1.03)

2. Primary Outcome: Impairment Rating Scale
Description: ADHD impairment - teacher rating. Average score ranges from 0.0 to 6.0 with higher scores indicating greater impairment.
Time Frame: Baseline (Fall), 3 Months (Winter), 6 Months (Spring) and 12 Months (First Grade Follow-up)
Measure: Mean (Standard Deviation); unit: Score on the scale
Arm/Group | School as Usual | Immediate Relative Age Effect Intervention | Delayed Relative Age Effect Intervention
Number analyzed (Participants) | 20 | 21 | 21
Score on the scale
  Fall (Baseline | 1.48 (2.01) | 2.25 (1.84) | 1.84 (1.71)
  Winter | 2.48 (2.15) | 2.43 (1.43) | 1.7 (1.66)
  Spring | 3.24 (2.30) | 2.19 (1.58) | 1.57 (1.55)
  Fall (First Grade Follow-up) | 2.22 (2.40) | 2.44 (2.06) | 1.86 (1.94)

3. Primary Outcome: Student Behavior Teacher Response Observation Code
Description: Number of disruptive behaviors; higher counts equal the presence of more classroom rule violations
Time Frame: Baseline (Fall), 3 Months (Winter), 6 Months (Spring) and 12 Months (First Grade Follow-up)
Measure: Mean (Standard Deviation); unit: Frequency count of behaviors
Arm/Group | School as Usual | Immediate Relative Age Effect Intervention | Delayed Relative Age Effect Intervention
Number analyzed (Participants) | 20 | 21 | 21
Frequency count of behaviors
  Fall (Baseline | 5 (4.27) | 5.67 (6.2) | 7 (6.7)
  Winter | 5.56 (8.12) | 5.21 (7.77) | 5.75 (4.9)
  Spring | 4.22 (4.02) | 4.36 (5.51) | 4.17 (3.74)
  First grade follow-up (Fall) | 3 (2.39) | 3.88 (3.74) | 2.6 (3.53)

4. Primary Outcome: Academic Performance Rating Scale
Description: Teacher rating of academic productivity. Average scores range from 1.0 to 5.0 with lower scores indicating academic underperformance.
Time Frame: Baseline (Fall), 3 Months (Winter), 6 Months (Spring) and 12 Months (First Grade Follow-up)
Measure: Mean (Standard Deviation); unit: Score on the scale
Arm/Group | School as Usual | Immediate Relative Age Effect Intervention | Delayed Relative Age Effect Intervention
Number analyzed (Participants) | 20 | 21 | 21
Score on the scale
  Fall (Baseline) | 3.51 (.83) | 3.22 (.97) | 3.36 (.97)
  Winter | 3.17 (.55) | 3.36 (.83) | 3.34 (.94)
  Spring | 3.15 (1.03) | 3.5 (.81) | 3.49 (.84)
  First Grade Follow-up (Fall) | 3.7 (.87) | 3.49 (.8) | 3.01 (1.09)

5. Other Pre Specified Outcome: Number of Children Who Were Referred to Special Education
Description: Dichotomous parent rating of yes or no for referral for special education at the end of kindergarten
Time Frame: Collected at the end of the kindergarten school year, approximately 10 months from the start of study procedures.
Measure: Count of Participants; unit: Participants
Arm/Group | School as Usual | Immediate Relative Age Effect Intervention | Delayed Relative Age Effect Intervention
Number analyzed (Participants) | 20 | 21 | 21
Participants | 1 | 2 | 3

6. Other Pre Specified Outcome: Number of Children Who Were Prescribed Stimulant Medication
Description: Dichotomous parent rating of yes or no for initiation of stimulant medication at the end of kindergarten
Time Frame: Collected at the end of the kindergarten school year, approximately 10 months from the start of study procedures.
Measure: Count of Participants; unit: Participants
Arm/Group | School as Usual | Immediate Relative Age Effect Intervention | Delayed Relative Age Effect Intervention
Number analyzed (Participants) | 20 | 21 | 21
Participants | 0 | 0 | 2

7. Other Pre Specified Outcome: Number of Children Who Were Retained in Kindergarten
Description: Dichotomous parent rating of yes or no for retained in kindergarten at the end of kindergarten
Time Frame: Collected at the end of the kindergarten school year, approximately 10 months from the start of study procedures.
Measure: Count of Participants; unit: Participants
Arm/Group | School as Usual | Immediate Relative Age Effect Intervention | Delayed Relative Age Effect Intervention
Number analyzed (Participants) | 20 | 21 | 21
Participants | 0 | 3 | 0

ADVERSE EVENTS:
Time Frame: 1 year, three months
Arm/Group | School as Usual | Immediate Relative Age Effect Intervention | Delayed Relative Age Effect Intervention
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT05142826/Prot_SAP_000.pdf